CLINICAL TRIAL: NCT02894164
Title: Evaluating the Role of Cystatin C and Creatinine as Markers of Renal Recovery in Critically Ill Patients After Acute Kidney Injury.
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Claire Rimes-Stigare, Doctor, Karolinska Institutet
Other Study IDs: CysCr1
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Acute Kidney Injury; Chronic Kidney Disease; Acute Kidney Disease
Keywords: Cystatin C; Creatinine; Glomerular Filtration Rate
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
This is a cohort study in which patients who survive Acute Kidney Injury (AKI) during intensive care unit (ICU) admission are recalled at 3-6 months and renal function tests are performed.

The purpose of the study is describe renal function in AKI survivors at follow-up.

Additional aims are to determine how well admission values of renal function markers perform as predictors of renal function at follow-up and whether estimates of renal function at follow-up differ depending on which renal function marker is used.

DETAILED DESCRIPTION:
Type of study: Cohort study with prospectively collected clinical data cross-matched with local & national databases.

Source population: Patients suffering from AKI on a mixed intensive care unit, at the Karolinska University Hospital, Solna.

Setting: Single centre, Central Intensive Care unit Karolinska University hospital, Solna, Stockholm from September 2008 and May 2011.

Exposure: AKI on ICU and grade of AKI according to the RIFLE criteria Intervention: none

Outcome: Renal function 3 months after ICU discharge according to creatinine and Cystatin C measurements.

Parameters: Co-morbidities, ICU diagnoses, disease severity score, daily physiological and laboratory parameters, medications administered, interventions RRT (Renal replacement therapy), mechanical intervention, inotropes, surgery.

Data is crossmatched with national registries including the Swedish cause of death register (to obtain dates of death), the Swedish renal register (to obtain details of patients receiving chronic dialysis and with pre-existing Chronic Kidney Disease (CKD) diagnoses. Data is also cross matched with a large local ICU register (Clinisoft) to obtain physiological parameters& intervention details. Clinisoft is also used to obtain risk of death for all ICU patients and all AKI patients (from the source population). Ethical approval has been granted by Stockholm Regional ethical review body (2008-408-32 2008/443-31/1-3, 2010/1780-31-2, 2011-408-32 and 2016-1801-32).

Aims:

1. Describe the incidence of renal dysfunction in terms of Glomerular filtration rate (GFR) under 60ml/min/173m² at 3-6 months follow-up after AKI. According to serum Cystatin C and Creatinine values.
2. Describe the incidence of Acute Kidney Disease (AKD) at 3 month follow-up.
3. Produce a predictive model using comorbidities and admission data to CKD (Chronic Kidney Disease) and AKD 3-6 after AKI in intensive care patients.
4. Examine how estimated GFR using creatinine and Cystatin C differ from measured Iohexol GFR at 6 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults treated on Intensive care with AKI (RIFLE criteria)
* Survival 3 months after discharge.
* Admission during September 2008-May 2011

Exclusion Criteria:

* Under 18 years
* Unable to give consent.
* Admission during a time when study staff not working.
* Death before 3 month follow-up
* No Swedish personal identification number

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the central intensive care unit at Karolinska University hospital, who suffered from AKI during the period September 2008 until May 2011.
Sampling Method: Non-Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Renal function | 3-9 months
  Renal function as defined by estimated glomerular filtration rate (eGFR)using seri Creatinine and Cystatin C at follow-up

SECONDARY OUTCOMES:
Mortality | 2 years
  Death as recorded in the swedish national death register.

CONTACTS AND LOCATIONS:
Overall Officials: Max Bell, PhD, Study Director — Karolinska Institutet; Johan Mårtensson, PhD, Principal Investigator — Karolinska Institutet; Claes-Roland Martling, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institute, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Data is anonymised and data regarding individuals will not be published.

REFERENCES:
- [Background] Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P; Acute Dialysis Quality Initiative workgroup. Acute renal failure - definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care. 2004 Aug;8(4):R204-12. doi: 10.1186/cc2872. Epub 2004 May 24. PMID 15312219